CLINICAL TRIAL: NCT01383590
Title: Identification of Potential Biomarkers of Peptide Immunotherapy. Part 1 - Proteomics Analysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RES-003
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Cat Allergy
Keywords: Cat allergy; Rhinoconjunctivitis; Immunotherapy; Cat-PAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cat-PAD (Experimental)
  Interventions: Biological: Cat-PAD

INTERVENTIONS:
Biological: Cat-PAD — Intradermal injection 1 x 4 administrations 4 weeks apart.

SUMMARY:
Cat allergy is an increasingly prevalent condition, affecting 10-15% of patients with allergic rhinoconjunctivitis. Cat-PAD is a novel synthetic, allergen derived peptide desensitizing vaccine currently being developed for the treatment of cat allergy.

At present, the efficacy of immunotherapy (peptide or otherwise) can only be established at the conclusion of therapy. The aim of this study is to identify changes in potential biomarkers after peptide immunotherapy that may be subsequently developed as biomarkers that equate with clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18-65 years
* A minimum 1-year documented history of rhinoconjunctivitis on exposure to cats.
* Positive skin prick test to cat allergen with a wheal diameter at least 3mm larger than that produced by the negative control.
* Regular exposure to a cat in their normal living or working circumstances throughout the course of the study.
* Minimum qualifying rhinoconjunctivitis symptom scores

Exclusion Criteria:

* History of asthma
* A history of anaphylaxis to cat allergen
* A history of allergen immunotherapy in the previous 10 years, or in the previous 3 years for pre-seasonal immunotherapy treatments
* A history of any significant disease or disorder (e.g. autoimmune, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment, severe atopic dermatitis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Identification of potential plasma biomarkers of response to peptide immunotherapy | 6 months following last treatment
  Blood samples derived from the study will be submitted for proteomics analyses aimed at the identification of one or more plasma proteins whose concentration over the course of the study varies in relation to the treatment administered. The outcome will be determined on the basis of measurements from samples collected over a period commencing prior to treatment and ending 6 months following treatment.

SECONDARY OUTCOMES:
Symptom scores for ocular and nasal symptoms | 4 weeks following treatment
Interleukin production and eosinophil level changes | 4 weeks following treatment
Functional genomic changes | 4 weeks following treatment
Changes in urine metabolomic profiles | 4 weeks following treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Neighbour H, Soliman M, Steacy LM, Hickey P, Forbes B, Larche M, Ellis AK. The Allergic Rhinitis Clinical Investigator Collaborative (AR-CIC): verification of nasal allergen challenge procedures in a study utilizing an investigational immunotherapy for cat allergy. Clin Transl Allergy. 2018 Apr 12;8:15. doi: 10.1186/s13601-018-0198-7. eCollection 2018. PMID 29682277